CLINICAL TRIAL: NCT02964208
Title: AMPLATZER™ LAA Occluder Post Approval Study
Brief Title: AMPLATZER™ LAA Occluder Post Approval Study (PAS)
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM-CIP-10122
Record Dates: First submitted 2016-10-06; First posted 2016-11-16 (Estimated); Results first posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Atrial Fibrillation; Thromboembolism; Stroke
Keywords: Atrial Fibrillation; Stroke; Left Atrial Appendage; Cardiac Plug; Amulet; Thromboembolism
MeSH Terms: conditions — Atrial Fibrillation; Thromboembolism; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- LAA Occluder PAS: Subjects who were treated with AMPLATZER LAA Occluders will be included.
  Interventions: Device: AMPLATZER™ LAA Occluder

INTERVENTIONS:
Device: AMPLATZER™ LAA Occluder — The AMPLATZER™ LAA Occluder is intended to prevent thrombus embolization from the left atrial appendage (LAA) in patients who have nonvalvular Atrial Fibrillation (AF). It may be considered for use in patients who have a high risk of stroke and bleeding and are deemed by their physician to have an appropriate rationale to seek a non-pharmacologic alternative to long term anticoagulants.
  Other Names: AMPLATZER™ Cardiac Plug™; AMPLATZER™ Amulet™

SUMMARY:
The aim of this multicenter, non-randomized observational post-approval is to compile real world outcome data on the use of an AMPLATZER LAA Occluder in subjects with non-valvular atrial fibrillation (NVAF). The AMPLATZER LAA Occluders is a transcatheter, self-expanding nitinol device intended for use in preventing thrombus embolization from the LAA.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Documented history of nonvalvular atrial fibrillation
* Subjects in whom an AMPLATZER LAA Occluder device is intended to be implanted or Subjects who underwent an AMPLATZER LAA Occluder implant attempt after the device was approved in the applicable geography

Exclusion Criteria:

* Women of childbearing potential who are, or plan to become, pregnant during the time of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population will include participants that are > 18 years old and diagnosed with NVAF.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Palmer, Study Director — Abbott
Locations (22):
- Instituto Cardiovascular de Rosario, Rosario, Santa Fe Province, Argentina
- Hôpital Civil Marie Curie, Lodelinsart, Hainaut, Belgium
- Canada (8):
  - Royal Columbian, New Westminster, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - CHUM, Montreal, Quebec
  - The Royal Victoria Hospital, Montreal, Quebec
- Chile (2):
  - Instituto Nacional del Torax, Providencia, Santiago Metropolitan
  - Hospital Clinico San Borja Arriarán, Santiago
- Germany (4):
  - Cardioangiologisches Centrum am Bethanien Krankenhaus, Frankfurt am Main, Hesse
  - St. Marien-Hospital-Bonn, Bonn, North Rhine-Westphalia
  - Segeberger Kliniken GmbH, Bad Segeberg, Schleswig-Holstein
  - Zentralklinik Bad Berka GmbH, Bad Berka, Thuringia
- Italy (3):
  - Azienda Ospedaliera Monaldi, Napoli, Campania
  - Ospedale San Giovanni Bosco, Torino, Piedmonte
  - Università degli Studi di Padova, Padua, Veneto
- Spain (3):
  - Hospital Universitario de Salamanca, Salamanca, Castille and León
  - Hospital Clinic I Provincial de Barcelona, Barcelona, Catalonia
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 520 patients were enrolled and underwent Amplatzer LAA Occluder implant attempt at 22 investigational sites between December 8, 2016 and July 2, 2020.
Period: Overall Study
Arm/Group | LAA Occluder PAS
Started | 520
Completed | 396
Not Completed | 124
Not completed — Death | 103
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 6
Not completed — Unsuccessful Procedure | 5
Not completed — Device Explant | 1
Not completed — Anatomical Heart Structure of the Patient; LAA Occluder Was Not Implanted; Heart Transplant | 3

BASELINE CHARACTERISTICS:
Arm/Group | LAA Occluder PAS
Number analyzed (Participants) | 520
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.90 (8.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 185
  Male | 335
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48
  Not Hispanic or Latino | 248
  Unknown or Not Reported | 224
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 16
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 0
  White | 303
  More than one race | 11
  Unknown or Not Reported | 187
Medical History [Count of Participants; unit: Participants]
  History of Major Bleeding | 392
  HAS-BLED score | 520
  History of TIA | 65
  History of Stroke | 160

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness Endpoint 1: Composite Rate of Stroke (Including Ischemic or Hemorrhagic), Systemic Embolism and Cardiovascular or Unexplained Death
Description: The occurrence of one or more the composite of stroke (including ischemic or hemorrhagic), systemic embolism, or cardiovascular or unexplained death at 24 months from the time of enrollment
Time Frame: Implant through 24 months
Population: The number of participants analyzed includes subjects for whom data were available at that time of analysis.
Measure: Number; unit: percentage of participants
Arm/Group | LAA Occluder PAS
Number analyzed (Participants) | 513
percentage of participants | 14.28

2. Primary Outcome: Primary Effectiveness Endpoint 2: Composite Rate of Ischemic Stroke or Systemic Embolism
Description: The occurrence of ischemic stroke or systemic embolism at 24 months from the time of enrollment
Time Frame: Implant through 24 months
Population: The number of participants analyzed includes subjects for whom data were available at that time of analysis.
Measure: Number; unit: percentage of participants
Arm/Group | LAA Occluder PAS
Number analyzed (Participants) | 513
percentage of participants | 4.41

3. Primary Outcome: Primary Safety Endpoint: Number of Subjects With All Cause Death, Ischemic Stroke, Systemic Embolism, or Device or Procedure-Related Events Requiring Open Cardiac Surgery or Major Endovascular Repair
Description: The occurrence of one of the following events between the time of implant and within 7 days of the procedure or by hospital discharge, whichever is later: all-cause death, ischemic stroke, systemic embolism, or device or procedure-related events requiring open cardiac surgery or major endovascular repair
Time Frame: Implant through 7 days
Population: The number of participants analyzed includes subjects for whom data were available at that time of analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | LAA Occluder PAS
Number analyzed (Participants) | 520
Participants | 3

4. Secondary Outcome: Comparison of the Relative Risk Decrease Of Observed Rate of Ischemic Stroke at 24 Months With the CHA2DS2-VASc Predicted Rate for the Implant Population
Description: The secondary endpoint comparing the observed rate of ischemic stroke at 24 months with the congestive heart failure, hypertension, age ≥ 75 years, diabetes mellitus, stroke or transient ischemic attack (TIA), vascular disease, age 65 to 74 years, sex category (CHA2DS2-VASc) score predicted rate for the implant population. The following calculation was used to calculate the Relative Risk Decrease: (Predicted Rate minus Observed Rate) divided by Predicted Rate = Relative Risk Decrease.
Time Frame: Implant through 24 months
Population: The number of participants analyzed includes subjects for whom data were available at that time of analysis.
Measure: Number; unit: percent change in the rate
Arm/Group | LAA Occluder PAS
Number analyzed (Participants) | 520
percent change in the rate | -70

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | LAA Occluder PAS
All-Cause Mortality (participants affected / at risk) | 103/520
Serious Adverse Events (participants affected / at risk) | 201/520
Other Adverse Events (participants affected / at risk) | 3/520
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LAA Occluder PAS (N=520)
Anemias (Blood and lymphatic system disorders) | 17
Iron-Deficiency Anemia (Blood and lymphatic system disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 3
Cardiac Arrest (Cardiac disorders) | 6
Cardiomyopathy (Cardiac disorders) | 2
Congestive Heart Failure (Cardiac disorders) | 7
Decompensated Heart Failure (Cardiac disorders) | 2
Heart Failure (Cardiac disorders) | 8
Mitral Valve Regurgitation/Mitral Insufficiency (Cardiac disorders) | 2
Myocardial Infarction (Cardiac disorders) | 3
Pericardial Effusion (Cardiac disorders) | 4
Pericardial Tamponade (Cardiac disorders) | 11
Pericarditis (Cardiac disorders) | 4
Persistent Atrial Fibrillation (Cardiac disorders) | 1
Sinus Bradycardia/Sinus Bradycardia (Cardiac Arrhythmia) (Cardiac disorders) | 1
Thrombus (Cardiac disorders) | 2
Retinal Hemorrhage (Eye disorders) | 1
Bowel Obstruction (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Gastrointestinal Bleeding (Gastrointestinal disorders) | 35
Ascites (General disorders) | 1
Change in Gait (General disorders) | 1
Dizziness (General disorders) | 1
Failure to Thrive (General disorders) | 1
Multiple Organ Failure (General disorders) | 5
Other (General disorders) | 10
Hepatic and Biliary Disorders (Hepatobiliary disorders) | 1
Pancreatic Cancer (Hepatobiliary disorders) | 1
Acute Bacterial Endocarditis (ABE) (Infections and infestations) | 1
Acute Peritonitis (Infections and infestations) | 1
Aspiration Pneumonia/Necrotizing Pneumonia/Aspiration of Vomitus (Infections and infestations) | 3
Chlamydial Pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 6
Pneumonia Caused By Gram-Negative Bacilli (Infections and infestations) | 1
Sepsis (Infections and infestations) | 9
Septicemia (Infections and infestations) | 1
Urinary Tract Infections (Infections and infestations) | 1
Viral Syndrome (Infections and infestations) | 1
Closed Head Injury (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hip Fracture (Injury, poisoning and procedural complications) | 2
Trauma (Injury, poisoning and procedural complications) | 2
Abnormal Lab Value (Investigations) | 1
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Acute Subdural Hematoma (Nervous system disorders) | 1
Delirium (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 3
Incidental Finding of Stroke (Nervous system disorders) | 1
Intracerebral Haemorrhage (Nervous system disorders) | 9
Ischemic Stroke (Nervous system disorders) | 17
Myoclonus (Nervous system disorders) | 1
Paresthesia/Paraesthesia (Nervous system disorders) | 1
Seizure/Convulsions/Epilepsy (Nervous system disorders) | 4
Stroke (Nervous system disorders) | 1
Transient Ischemic Attack (TIA) (Nervous system disorders) | 4
Vertigo (Nervous system disorders) | 1
Device Migration (Product Issues) | 1
Thrombus on Device (Product Issues) | 3
Acute Kidney Injury (Renal and urinary disorders) | 1
Acute Renal Failure (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 5
Renal Insufficiency (Renal and urinary disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Idiopathic Interstitial Lung Diseases (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 7
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 8
Hemarthrosis (Skin and subcutaneous tissue disorders) | 1
Seroma (Skin and subcutaneous tissue disorders) | 1
Arterial Hypertension/Hypertension (Vascular disorders) | 1
Bleeding (Vascular disorders) | 3
Carotid Aneurysm (Vascular disorders) | 1
Deep Vein/Venous Thrombosis (Vascular disorders) | 1
Hematoma (Vascular disorders) | 7
Hemorrhage (Vascular disorders) | 1
Hypertensive Crisis (Vascular disorders) | 1
Perforation of Vessel (Vascular disorders) | 2
Peripheral Arterial Occlusion (Vascular disorders) | 2
Syncope (Vascular disorders) | 1
VASC Bleeding (Vascular disorders) | 2
VASC Pseudoaneurysm (Vascular disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LAA Occluder PAS (N=520)
Thrombus on Device (Product Issues) | 1
Transient Ischemic Attack (TIA) (Nervous system disorders) | 1
Unstable Angina (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/08/NCT02964208/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/08/NCT02964208/SAP_001.pdf